CLINICAL TRIAL: NCT06716736
Title: Socket Preservation Using Autogenous Particulate Dentin in Combination With Liquid Platelet-rich Fibrin Versus Bone Allografts and Collagen Cones After Surgical Extraction of Impacted Lower Third Molar
Brief Title: Socket Preservation After Surgical Extraction of Impacted Lower Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Mohamed (Other)
Responsible Party: Sponsor-Investigator, Wael Mohamed, Professor of Oral and Maxillofacial Surgery, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A08061222
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Socket Preservation
Keywords: socket preservation; dentine graft
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- socket preservation with dentine graft mixed with liquid platelet rich fibrin (sticky tooth) (Active Comparator): socket preservation with dentine graft mixed with liquid platelet rich fibrin (sticky tooth) after surgical extraction of horizontally impacted lower wisdom
  Interventions: Biological: socket preservation using dentine graft mixed with i-PRF
- socket preservation with bone allograft (Active Comparator): socket preservation with bone allograft after surgical extraction of horizontally impacted lower wisdom
  Interventions: Biological: socket preservation using bone allograft
- socket preservation with collagen cone (Active Comparator): socket preservation with collagen cone after surgical extraction of horizontally impacted lower wisdom
  Interventions: Biological: socket preservation using collagen cone

INTERVENTIONS:
Biological: socket preservation using dentine graft mixed with i-PRF — surgical extraction of horizontally impacted third molar , placement of dentin graft mixed with i-PRF inside the socket , suturing
  Arms: socket preservation with dentine graft mixed with liquid platelet rich fibrin (sticky tooth)
Biological: socket preservation using bone allograft — surgical extraction of horizontally impacted third molar , placement of bone allograft inside the socket , suturing
  Arms: socket preservation with bone allograft
Biological: socket preservation using collagen cone — surgical extraction of horizontally impacted third molar , placement of collagen cone inside the socket , suturing
  Arms: socket preservation with collagen cone

SUMMARY:
The aim of this study will be to evaluate socket preservation using autogenous particulate dentin in combination with liquid platelet-rich fibrin versus bone allografts and collagen cone after surgical extraction of the horizontally impacted lower third molar

DETAILED DESCRIPTION:
The aim of this study will be to evaluate socket preservation using autogenous particulate dentin in combination with liquid platelet-rich fibrin (sticky tooth) versus bone allografts and collagen cone after surgical extraction of the horizontally impacted lower third molar

ELIGIBILITY:
Inclusion Criteria:

1. Fresh extracted socket of horizontally impacted mandibular third molar
2. Co-operative patients willing to complete the follow-up periods.
3. Patients age from 18-35 years.
4. Good oral hygiene.

Exclusion Criteria:

1. Any pathological condition at the site of surgery.
2. Patients with systemic diseases that contra-indicate the surgical procedure such as uncontrolled diabetes mellitus, bleeding disorders, serious osseous disorders and mental disorders.
3. Smokers .
4. Pregnancy.

   -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
bone resorption distal to second molar | 3 months after extraction
  by measuring bone level immediate and 3 months after extraction on CBCT

SECONDARY OUTCOMES:
bone density | 3 months after extraction
  using CBCT 3 month after extraction
edema | 4 days after extraction
  by measuring distance between predetermined anatomical landmarks:
  * Mandibular angle and canthus of the eye.
  * Mandibular angle and corner of the mouth.
  * Mandibular angle and tragus.
  * Mandibular angle and pogonion.
pain after surgical extraction | 4 days after extraction
  using numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wael M Ahmed, PHD, Principal Investigator — mansoura uniersity
Locations (1):
- Mansoura University, Al Mansurah, Eldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No